CLINICAL TRIAL: NCT06072612
Title: Randomized, Open-Label Study of the Bria-IMT Regimen and Check Point Inhibitor vs Physicians' Choice in Advanced Metastatic Breast Cancer.
Brief Title: Study of the Bria-IMT Regimen and CPI vs Physicians' Choice in Advanced Metastatic Breast Cancer.
Acronym: BRIA-ABC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BriaCell Therapeutics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC-IMT-04
Record Dates: First submitted 2023-09-25; First posted 2023-10-10 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Metastatic Breast Cancer; Breast Neoplasm; Breast Cancer Metastatic; End Stage Cancer
Keywords: Breast; metastatic; advanced; cancer; late line
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Bria-IMT Regimen + CPI (Experimental): The Bria-IMT regimen:
  Day -2 or -3 Cyclophosphamide 300mg/m2 Day 0 SV-BR-1-GM given intradermally divided into 4 inoculations Day 1-3 CPI infusion plus interferon administered intra-dermally within each SV-BR-1-GM inoculation site
  Interventions: Biological: SV-BR-1-GM; Drug: Cyclophosphamide; Drug: Interferon infiltration of the inoculation site; Drug: Retifanlimab
- Treatment of Physician's Choice (Active Comparator): TPC consists of eribulin, carboplatin, capecitabine, gemcitabine, vinorelbine or taxanes in accordance with the investigators' and institutional standard of care. The specific details of the selected regimen must include every detail of administration including frequency, sequencing (for multi-agent regimens), duration of infusion or oral administration, planned dose, dose prescribed, dose administered, dose adjustments after initial prescription or start of TPC treatment, and any other change in TPC from its initial election prior to randomization.
  Interventions: Drug: Treatment of Physician's Choice
- Bria-IMT Regimen Alone (Experimental): The Bria-IMT regimen:
  Day -2 or -3 Cyclophosphamide 300mg/m2 Day 0 SV-BR-1-GM given intradermally divided into 4 inoculations Day 1-3 CPI infusion plus interferon administered intra-dermally within each SV-BR-1-GM inoculation site
  Interventions: Biological: SV-BR-1-GM; Drug: Cyclophosphamide; Drug: Interferon infiltration of the inoculation site

INTERVENTIONS:
Biological: SV-BR-1-GM — SV-BR-1-GM is an experimental, allogeneic, whole cell breast tumor cell line stably transfected with the CSF2 gene (encoding GM-CSF) to secrete GM-CSF in vivo to consequently augment dendritic cell activity
  Other Names: Part of the Bria-IMT regimen
  Arms: Bria-IMT Regimen + CPI; Bria-IMT Regimen Alone
Drug: Cyclophosphamide — Cyclophosphamide is an alkylating agent with indications for treatment of malignant diseases including breast cancer. Cyclophosphamide (Cytoxan) 300 mg/m2 I.V., single dose, will be given to patients assigned to the SV-BR-1-GM. Cyclophosphamide will be administered 2-3 days prior to SV-BR-1-GM inoculations.
  Arms: Bria-IMT Regimen + CPI; Bria-IMT Regimen Alone
Drug: Interferon infiltration of the inoculation site — Interferon is a cytokine released by cells to regulate immune responses to viral infections. For this study, 0.1 mcg Pegasys per injection site (x 4 injection sites) will be administered.
  Arms: Bria-IMT Regimen + CPI; Bria-IMT Regimen Alone
Drug: Retifanlimab — Retifanlimab is a checkpoint inhibitor. A total dose of 375mg will be administered at first cycle on or about day +2 (+/-1d). In all other cycles, Retifanlimab is permitted to be administered between Day -2/-3 to Day 2±1 of the cycle based on the convenience of the patients and the clinical sites. However once the timing of the CPI is chosen for C1, it must be given on the same day thereafter throughout the trial.
  Arms: Bria-IMT Regimen + CPI
Drug: Treatment of Physician's Choice — Patients in the TPC arm of the study will be treated with one or a combination of the following: carboplatin, taxanes, capecitabine, gemcitabine, vinorelbine or eribulin in accordance with the investigators and institutional standard of care. For HER2+ patients, a HER2-targeted agent of the physician's choice can be part of TPC.
  Arms: Treatment of Physician's Choice

SUMMARY:
This is a multicenter randomized, open label study to evaluate overall survival with the Bria-IMT regimen in combination with Checkpoint Inhibitor [Retifanlimab], versus Treatment of Patients'/Physicians' Choice (TPC) in advanced metastatic or locally recurrent breast cancer (aMBC) patients with no approved alternative therapies available.

DETAILED DESCRIPTION:
This is a multicenter randomized, open label study to evaluate overall survival with the Bria-IMT regimen in combination with Checkpoint Inhibitor [Retifanlimab], versus Treatment of Patients'/Physicians' Choice (TPC) in advanced metastatic or locally recurrent breast cancer (aMBC) patients with no approved alternative therapies available. A secondary objective will be to evaluate the activity of the Bria-IMT regimen alone in comparison with the Bria-IMT regimen in combination with CPI.

Initial randomization will be 1:1:1 to the Bria-IMT regimen + CPI (combination therapy), TPC, and the Bria-IMT regimen alone (monotherapy). After the first 150 patients have enrolled in the study, the monotherapy arm will be discontinued and patients allowed to cross over to the combination therapy if needed. Randomization will continue 1:1 between the combination therapy vs TPC.

For the Bria regimen +/- CPI arms, treatment cycles occur every 3 weeks. TPC cycle details will be according to the site's SOC. In the absence of progressive disease or major safety issues, the patient will continue with therapy cycles, with imaging assessment every 6 weeks x2 then every 8 weeks thereafter.

The Bria-IMT regimen includes:

Day -2 or -3 Cyclophosphamide 300mg/m2 Day 0 SV-BR-1-GM given intradermally divided into 4 inoculations Day 1-3 CPI infusion plus interferon intra-dermally within each Bria-IMT inoculation site

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥ 18 years of age.
2. Have signed informed consent.
3. Have histological confirmation of breast cancer with either locally recurrent unresectable and/or metastatic lesions, and have failed prior therapy:

   * Patients with persistent disease and local recurrence must not be amenable to local treatment.
   * For patients with metastatic disease, late-stage MBC with no meaningful alternative therapies available and the following class specific treatment histories:

     1. Human epidermal growth factor 2 (HER2) positive must be previously treated with at least 3 regimens containing at least two anti-HER2 and at least one chemotherapy containing regimen.
     2. Estrogen receptor (ER), progesterone receptor (PR) positive tumors: must be refractory to hormonal therapy demonstrated by progression on at least 2 hormonal agents in 2 separate lines of hormone directed therapy.
     3. Triple Negative tumors: Must have exhausted all curative intent therapies including at least 2 prior chemotherapy regimens, which can include regimens in neoadjuvant and adjuvant settings.
     4. Cancers with known germline or genomic actionable targets, e.g. g/mBRCA, must have been treated with all tumor directed indicated treatment e.g. PARPi, if tolerated.
     5. HER2 low patients, in addition to the appropriate therapies based on ER/PR status and germline or genomic actionable targets, must also have received at least one HER2-targeted agent approved for treatment of HER2 low patients.
     6. HER2 negative tumors must be refractory to hormonal therapy (if indicated) and previously treated with at least 2 chemotherapy regimens.
     7. Patients with new or progressive breast cancer metastatic to the brain will be eligible provided:

        * The brain metastases must be clinically stable (without evidence of progressive disease by imaging for at least 4 weeks prior to first dose)
        * There is no need for steroids and patients have not had steroids for at least 2 weeks prior to the first dose
        * Tumor is not impinging on Middle Cerebral Artery/speech-motor strip
        * If surgically debulked, must be healed with at least 3 weeks since surgery prior to the first dose
4. Has expected survival of at least 4 months.
5. ECOG performance status of 0, 1 or 2

Exclusion Criteria:

1. Concurrent or recent chemotherapy, immunotherapy or major surgery within 21 days prior to the first dose.
2. Radiotherapy within 14 days of the first dose of study treatment.
3. Toxicity of prior therapy that has not recovered to ≤ Grade 1 or baseline (with the exception of any grade of alopecia and anemia not requiring transfusion support).
4. Any toxicity to prior CPI that was grade 3 or higher unless it has been successfully treated (e.g. hypothyroidism or hypopituitarism treated with replacement therapy), .
5. Toxicity to prior CPI that has not resolved to grade 1 or less except for stable asymptomatic endocrinopathies.
6. History of clinical hypersensitivity to the designated therapy as specified in the protocol, including the proposed TPC, beef, or to any components used in the preparation of SV- BR-1-GM.
7. History of hypersensitivity to any of the therapies proposed for treatment in this study.
8. Serum creatinine OR Measured OR calculated Creatinine Clearance (CrCl) (GFR can also be used in place of creatinine or CrCl) >2.0 × ULN or <30 mL/min for participants with creatinine levels >2.0 × institutional ULN.
9. Absolute granulocyte count <1000; platelets <80,000; hemoglobin ≤ 7 g/L.
10. Bilirubin ≥ 2 × ULN unless conjugated bilirubin ≤ ULN; alkaline phosphatase >5x upper limit of normal (ULN); ALT/AST >3x ULN. For patients with hepatic metastases, ALT/AST >5x ULN is exclusionary.
11. INR or PT or aPTT > 1.8 × ULN, unless the participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants.
12. Receiving any medication listed in the prohibited medication section of the protocol.
13. Proteinuria >2+ on urinalysis
14. A history or presence of an abnormal electrocardiogram (ECG) that, in the Investigator's opinion, is clinically meaningful. Screening corrected QT interval (QTc) interval >480 milliseconds is excluded (corrected by Fridericia or Bazett formula). In the event that a single QTc is >480 milliseconds, the participant may enroll if the average QTc for the 3 ECGs is <480 milliseconds.
15. New York Heart Association stage 3 or 4 cardiac disease.
16. A pericardial effusion of moderate severity or worse.
17. Symptomatic pleural effusion or ascites. A participant who is clinically stable following treatment for these conditions (including therapeutic thoraco- or paracentesis) is eligible.
18. Any woman of childbearing potential (i.e., has had a menstrual cycle within the past year and has not been surgically sterilized), unless she agrees to take appropriate precautions to avoid becoming pregnant during the study and has a negative serum pregnancy test within 7 days prior to starting treatment.
19. Men must have been sterile or, if they were potentially fertile/reproductively competent, should take appropriate precautions to avoid fathering a child for the duration of the study.
20. Women who are pregnant or nursing.
21. Known additional malignancy that is progressing or requires active treatment, or history of other malignancy within 2 years of study entry with the exception of cured basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive or indolent malignancy, or cancers from which the participant has been disease-free for > 1 year, after treatment with curative intent.
22. Patients who have uncontrolled HIV or have clinical or laboratory features indicative of AIDS.
23. Have a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (doses exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.
24. Have an active autoimmune disease that has required systemic treatment in past year (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is allowed.
25. Known active HAV, HBV, or HCV infection, as defined by elevated transaminases with the following serology: positivity for HAV IgM antibody, anti-HCV, anti-HBc IgG or IgM, or HBsAg (in the absence of prior immunization).
26. Active infections requiring systemic therapy within the past 14 days.
27. Patients with severe psychiatric disease (e.g., schizophrenia, bipolar, or borderline personality disorder) or other clinically progressive major medical problems, unless approved by the Investigator in consultation with the Medical Monitor.
28. Has received a live vaccine within 28 days of the first dose of study drug.
29. Patients may not be on a concurrent clinical trial, unless approved by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Up to 60 months
  To evaluate the effect of the Bria-IMT regimen in combination with Check Point Inhibitor (CPI) on overall survival (OS) compared to treatment of physician's choice (TPC) chemotherapy in patients with metastatic breast cancer with no approved alternative therapies available as per the Inclusion criteria.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 60 months
  To evaluate the effect of the Bria-IMT regimen with CPI on progression-free survival (PFS)
  • To assess the single agent activity of the Bria-IMT regimen in the sample cohort using PFS, ORR, and CBR
Clinical Benefit Rate (CBR) | Up to 60 months
  To evaluate the efficacy of the Bria-IMT regimen with CPI using Clinical Benefit Rate (CBR)
Overall response rate (ORR) | Up to 60 months
  To evaluate the efficacy of the Bria-IMT regimen with CPI using best overall response rate (ORR)
Quality of life (QoL) | Up to 60 months
  To compare the effect of the Bria-IMT regimen with CPI on quality of life (QoL) including time without symptoms and time without toxicities (TWiST) adjusted for time on study.
CNS Event free survival (EFS) | Up to 60 months
  CNS event free survival for subjects with and without known CNS metastases at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Del Priore, MD MPH, Study Director — BriaCell Therapeutics
Locations (77):
- United States (77):
  - Mayo Clinic-Comprehensive Cancer Center-Breast Clinic, Phoenix, Arizona
  - University of Arizona-Cancer Center, Tucson, Arizona
  - Los Angeles cancer Network_Anaheim, Anaheim, California
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Cedars-Sinai Cancer Beverly Hills, Beverly Hills, California
  - Los Angeles Cancer Network_Corona, Corona, California
  - Los Angeles cancer Network_Fountain Vallley, Fountain Valley, California
  - Los Angeles Cancer Network_Glendale, Glendale, California
  - Hoag Hospital Center, Irvine, California
  - Hoag Hospital Irvine, Irvine, California
  - Los Angeles Cancer Network, Los Angeles, California
  - Cedars-Sinai Cancer at Cedars-Sinai Medical Facility, Los Angeles, California
  - Los Angeles Cancer Network_Century City, Los Angeles, California
  - UCLA-Hematology/Oncology Medical Plaza, Los Angeles, California
  - UCLA-Hematology/Oncology_LA 2, Los Angeles, California
  - UCLA-Hematology/Oncology_LA, Los Angeles, California
  - Los Angeles Cancer Network_Pasadena, Pasadena, California
  - Los Angeles cancer Network_Riverside, Riverside, California
  - UC San Diego, San Diego, California
  - St. John's Cancer Center, Santa Monica, California
  - UCLA-Department of Medicine Hematology/Oncology-Parkside, Santa Monica, California
  - UCLA-Hetamtology/Oncology_S Monica, Santa Monica, California
  - Torrance Memorial Cancer Center, Torrance, California
  - Los Angeles Cancer Network_Valley Pres, Van Nuys, California
  - Cedars-Sinai Breast Health Services Building, West Hollywood, California
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - University of Miami _SCCC - Aventura, Aventura, Florida
  - University of Miami-SCCC-Lennar, Coral Gables, Florida
  - University of Miami_SCCC-Coral Springs, Coral Springs, Florida
  - University of Miami Hospital and Clinics - Deerfield Beach, Deerfield Beach, Florida
  - University of Miami_SCCC-Hollywood, Hollywood, Florida
  - Mayo Clinic Florida-Comprehensive Cancer Center, Jacksonville, Florida
  - University Of Miami-SCCC-Miami, Miami, Florida
  - University of Miami_SCCC - Kendall, Miami, Florida
  - Advent Health - Orlando, Orlando, Florida
  - University of Miami-SCCC-Plantation, Plantation, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Southern Illinois University-Simmons, Springfield, Illinois
  - Carle Foundation Cancer Institute-Urbana, Urbana, Illinois
  - Northwest Cancer Center, Dyer, Indiana
  - AMR Kansas City Oncology, Kansas City, Kansas
  - Care Access-Marrero, Marrero, Louisiana
  - The Center for Cancer and Blood Disorders a division of American Oncology Partners, P.A., Bethesda, Maryland
  - Mayo Clinic-Comprehensive Cancer Center-Breast Clinic, Rochester, Minnesota
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hunterdon Medical Center, Flemington, New Jersey
  - New York Cancer and Blood Specialists_North Shore Hematology Oncology Assocaites P.C. (Babylon), Babylon, New York
  - New York Cancer and Blood Specialists_North Shore Hematology Oncology Assocaites P.C.(New Hyde Park), New Hyde Park, New York
  - Manhattan Hematology /Oncology Associates, New York, New York
  - New York Cancer and Blood Specialists_North Shore Hematology Oncology Assocaites P.C (NY), New York, New York
  - New York Cancers & Blood Specialists_North Shore Hematology Oncology Assocaites P.C (Patchogue), Patchogue, New York
  - New York Cancer and Blood Specialists_North Shore Hematology Oncology Assocaites P.C. (Port Jefferson Station2), Port Jefferson Station, New York
  - New York Cancer and Blood Specialists_North Shore Hematology Oncology Assocaites P.C.(Port Jefferson Station1), Port Jefferson Station, New York
  - New York Cancers & Blood Specialists, Port Jefferson Station, New York
  - New York Cancer and Blood Specialists_North Shore Hematology Oncology Assocaites P.C. (Riverhead), Riverhead, New York
  - New York Cancer and Blood Specialists_North Shore Hematology Oncology Assocaites P.C (Brox), The Bronx, New York
  - Gabrail Cancer & Research Center, Canton, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Mary Crowley Cancer Research, Dallas, Texas
  - DHR Health Oncology Institute, Edinburg, Texas
  - Texas Oncology - Fredericksburg, Fredericksburg, Texas
  - Texas Oncology - Harlingen, Harlingen, Texas
  - Texas Oncology McAllen, McAllen, Texas
  - Texas Oncology, New Braunfels, New Braunfels, Texas
  - Texas Oncology-San Antonio Cancer Care, San Antonio, Texas
  - Texas Oncology - San Antonio Northeast, San Antonio, Texas
  - Texas Oncology - San Antonio Stone Oak, San Antonio, Texas
  - Tranquil Clinical Research, Webster, Texas
  - Texas Oncology - Weslaco, Weslaco, Texas
  - Hematology-Oncology Associates of Fredericksburg, Inc, Fredericksburg, Virginia
  - Cancer Care Northwest-1 (601 S. Sherman), Spokane, Washington
  - Cancer Care Northwest_2 (605 E. Holland), Spokane, Washington
  - Cancer Care Northwest, Spokane Valley, Washington
  - Sheboygan Cancer & Blood Specialists, Sheboygan, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor — https://briacell.com/
- See also: CRO — https://www.prevailinfoworks.com/